CLINICAL TRIAL: NCT03104166
Title: Modulation of Vascular Calcification in Chronic Dialysis Patients
Acronym: ModuVas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Daniel Zickler, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ModuVas
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Vascular Calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO (Experimental): Patients will be treated thrice weekly with Medium Cut-Off Dialysis membranes.
  Interventions: Device: Medium Cut-Off (MCO) dialysis membrane
- High-Flux (Active Comparator): Patients will be treated thrice weekly with High-Flux Dialysis membranes.
  Interventions: Device: High-Flux dialysis membrane

INTERVENTIONS:
Device: Medium Cut-Off (MCO) dialysis membrane — Patients will be treated with a CE-certified dialysis membrane that provide enhanced clearance for middle-sized molecules, call Medium Cut-Off membrane.
  Arms: MCO
Device: High-Flux dialysis membrane — Control: Patients will be treated with a CE-certified High-Flux dialysis membrane.
  Arms: High-Flux

SUMMARY:
50 patients will be randomized and treated with MCO or highflux dialysis for six months (24 weeks) after a run-in phase of 4 weeks Highflux treatment.

Serum samples will be drawn at baseline, after 4, 8 and 24 weeks.

Later, calcifiying vascular smooth muscle cells will be incubated with these serum samples and calcification will be assessed with Alkaline phosphatase and Alizarin staining.

Primary endpoint:

In vitro Calcification of coronary vascular smooth muscle cells (Alkaline Phosphatase/ WST8) after six months

Calcifiying vascular smooth muscle cells will be incubated with serum samples obtained after six months of MCO/HF dialysis and calcification will be assessed with Alkaline phosphatase and WST8.

Secondary Endpoints:

Aortic Pulse wave velocity after 6 months Calcification propensity after 6 months Physical activity level after 6 months

Cell culture: Incubation of VSMC with serum samples obtained after 6 months

* Alizarin staining/WST-8
* Measurement of calcification inhibitors Osteopontin and Matrix Gla Protein in Supernatants
* Apoptosis

The treatment regimen of the patients will not be altered, hence blood flow, dialysate flow as well as dialysis time will remain constant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years an older
* Chronic dialysis patients for at least 3 months

Exclusion Criteria:

* Serum albumin <32g/L at the last routine albumin measurement
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
In vitro Calcification of coronary vascular smooth muscle cells (Alkaline Phosphatase/ WST8) after six months | Six months
  Serum samples will be drawn at the beginning of the trial and after six months treatment with either High-Flux or Medium Cut-Off filters. Vascular smooth muscle cells will be incubated with thee serum samples and calcification will be assessed with Alkaline Phosphatase/ WST8

SECONDARY OUTCOMES:
Aortic Pulse wave velocity | Six months
  Aortic Pulse wave velocity will be determined using the Vicorder Device.
Calcification propensity | Six months
  Calcification propensity will be determined as described earlier. (PMID: 24179171)
Physical activity level | Six months
  Physical activity level will be monitored for one week before and after treatment using an activity tracker.
Cell culture: Incubation of VSMC with serum samples and assessment of • Alizarin staining/WST-8 • Measurement of calcification inhibitors Osteopontin and Matrix Gla Protein in Supernatants • Apoptosis | Six months
  Additional in vitro calcification parameters will be assessed after incubation of VSMC with patient serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Virchow, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No